CLINICAL TRIAL: NCT03983590
Title: Analgesia Nociception Index (ANI) for Pain and Anxiety Assessment in Palliative Care : a Pilot Study in University Hospital of Rennes
Brief Title: Anxiety, Pain et Analgesia Nociception Index (ANI) in Palliative Care
Acronym: ADA-Pallia
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3054_ADA-PALLIA
Record Dates: First submitted 2019-06-06; First posted 2019-06-12 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Pain; Anxiety; Palliative Care
Keywords: pain; anxiety; communicative; palliative care
MeSH Terms: conditions — Pain; Anxiety Disorders; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Visual Analogic Scale — VAS are collected in the first 24 hours after inclusion, 15 minutes, during and 15 minutes after the bed bath. Each time of collection are noted.

SUMMARY:
The main objective of this study is to evaluate the correlation between ANI and pain scores and the correlation of ANI and anxiety scores in communicative patients in palliative care.

The chosen event with a risk of pain and/or anxiety is the first bed bath after admission. The secondary objectives aim to identify ANI score thresholds which would be predictive of pain and/or anxiety and to figure out some individual factors influencing ANI scores.

DETAILED DESCRIPTION:
Pain and anxiety assessments are still challenges for palliative care teams. Anxiolytics and painkillers are the usual tools but sometimes the symptoms and so the drugs to deliver are difficult to distinguish. For patients with maintained communication abilities, pain self-assessment using Visual Analogic Scores are the gold standard. Could pain assessment be optimised thanks to ANI? ANI is used in anaesthesiology and intensive care. The ANI system is based on the analysis of intra-cardiac variability. Based as an electrocardiograph with two electrodes on the patient's chest, it measures the balance between sympathetic/parasympathetic tones leading to a pain score. This score is predictive of pain occurrence, leading to an early analgesic treatment and a better control of pain with less quantity of drugs. However, some studies reported that anxiety and emotions could influence ANI pain score.

To test this hypothesis in palliative care field, this study compares pain and anxiety VAS to ANI scores before, during and after the bed bath.

ELIGIBILITY:
Inclusion Criteria:

* admitted in palliative care

  -≥18 years old
* enough communication abilities to use VAS
* non opposition of the patient

Non-inclusion criteria :

* previous bed bath already provided to the patient in the palliative unit (anxiolytic and analgesic strategies already adapted limiting the risk of pain or anxiety and the power of the study )
* adult under legal protection (guardianship, trusteeship …)
* contraindication of ANI : respiratory rate < 10/min, non sinusal cardiac rythm, cardiotropic treatments
* behavioural disorders : agitation, confusion (Richmond scale score > ou = 1)
* alertness disorders : somnolence (Richmond scale score < ou = -1)
* no French speaking

Exclusion criteria:

* providing the bad bath is impossible
* secondary opposition of the patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have just been admitted in palliative care unit and who have communication abilities enough for pain and anxiety self-assessment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
correlation rate of ANI (Analgesia Nociception Index) scores and pain Visual Analogic Scale (VAS) scores at each measurement time. | VAS are collected in the first 24 hours after inclusion, 15 minutes, during and 15 minutes after the bed bath. Each time of collection are noted.
  ANI scores, pain VAS and anxiety VAS scores are the basic measures which will allow the needed calculations.
  Significant results will be :
  * the correlation rate of ANI (Analgesia Nociception Index) scores and pain Visual Analogic Scale (VAS) scores
  * the correlation rate of ANI scores and anxiety scores After a descriptive study of collected variables, the correlation rates between ANI scores and VAS scores will be calculated. Linear regression or mixt gamma will be used to assess the intra-individual variability (random effect). The effect of individual variables on the ANI scores will be tested (age, sex, diseases, medications) Considering 3 as the significant VAS threshold, ROC curves and Younden indice will be used to identify ANI scores leading to prediction of pain and/or anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume ROBERT, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre Hospitalier Universitaire de Rennes, Rennes, France